CLINICAL TRIAL: NCT03376542
Title: Cardiopulmonary Exercise Testing as an Outcome Predictor in Coronary Artery Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eduardo Tibirica, MD, PhD (Other Government)
Responsible Party: Sponsor-Investigator, Eduardo Tibirica, MD, PhD, Senior Researcher, National Institute of Cardiology, Laranjeiras, Brazil
Organization: National Institute of Cardiology, Laranjeiras, Brazil (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CAAE: 67629917.1.0000.5272
Record Dates: First submitted 2017-11-22; First posted 2017-12-18 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Coronary Artery Disease; Surgery--Complications
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: All patients included in the study will perform cardiopulmonary exercise testing prior to surgery
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiopulmonary exercise testing (Experimental): All patients included in the study will perform cardiopulmonary exercise testing prior to surgery
  Interventions: Diagnostic Test: Cardiopulmonary Exercise Testing

INTERVENTIONS:
Diagnostic Test: Cardiopulmonary Exercise Testing — Cardiopulmonary exercise testing on treadmill prior to coronary artery bypass grafting surgery

SUMMARY:
This is a prospective cohort study of patients undergoing coronary artery bypass graft surgery. Prior to surgery, participants will undergo submaximal cardiopulmonary exercise testing on a treadmill. Participants will be followed for one month after surgery to assess mortality and non fatal complications.

DETAILED DESCRIPTION:
Coronary artery bypass surgery (CABG) is a complex and expensive procedure with great potential for morbidity and mortality. Preoperative evaluation is of paramount importance to optimize results. There is much evidence about the benefits of the cardiopulmonary exercise testing (CPET) in the evaluation of preoperative risk in non-cardiac surgeries. Thus, it is important to evaluate the relationship between parameters obtained in the CPET and the outcomes after cardiac surgery, especially CABG.

This is a prospective cohort study in which participants undergo submaximal CEPT on a treadmill prior to CABG. Participants will be followed up for one month after surgery to assess mortality and non fatal complications. It is expected that poor cardiopulmonary fitness is related to worse outcomes in CABG, as already observed in other cardiac pathologies and in non-cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing coronary artery bypass grafting surgery at the National Institute of Cardiology, Ministry of Health, Rio de Jnaeiro, Brazil.

Exclusion Criteria:

* Angina CCS IV, heart failure NYHA IV, inability to walk on a treadmill, severe left main coronary artery lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Mortality after cardiac surgery | 30 days
  number of deaths during the first 30 days after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Tibiriça, MD, PhD, Study Chair — National Institute of Cardiology, Laranjeiras, Brazil
Locations (1):
- National Institute of Cardiology, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No